CLINICAL TRIAL: NCT01817140
Title: Assessment of Mandibular Bone Invasion With Magnetic Resonance Imaging (MRI) Using Sweep Imaging Fourier Transformation (SWIFT)
Brief Title: Assessment of Mandibular Bone Invasion With MRI Using SWIFT
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NM2012-06-06
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Oral Cancer
Keywords: oral cancer; mandibular invasion; SWIFT MRI
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patient MRI: Adult patients with possible maxillofacial and/or mandibular bone invasion with oral cancer or osteoradionecrosis who are scheduled for surgery. All eligible and consented participants will have MRI scans obtained using 3T and 4T magnets prior to their surgery.
- Normal MRI: Healthy adult volunteers recruited to test the comfort of the coil apparatus and to determine configurations which lead to satisfactory image acquisition.

SUMMARY:
The primary objective of this study is to improve the diagnostic accuracy and specificity of MRI in detecting the degree of bone involvement and invasion in oral cancer. The presence and degree of bone invasion determines the extent of surgery and has great effect on the morbidity of patients with oral cancer and bone/soft tissue tumors.

MRI scanning in 3 Tesla (3T) and 4Tesla (4T) MR magnet will be performed on up to 10 patients with possible maxillofacial and/or mandibular bone invasion. We will then compare the conventional imaging results of the patients with 3T and 4T MRI results and post operative pathology results.

DETAILED DESCRIPTION:
Unfortunately, detecting bone invasion and extension of bone involvement prior to surgery is often difficult with the currently available imaging techniques. MRI with high contrast resolution and the ability to perform multiplanar imaging plays an integral role in the delineation of tumoral involvement of the bone. Although MRI is an excellent tool in the assessment of bone invasion in carcinoma, its overestimation of cortical invasion and tumor extent to the bone marrow have been a diagnostic challenge, leading to false positive results. Like many of the musculoskeletal system tissues, cortical bone produces no signal with conventional MRI techniques, limiting the characterization of image contrast and differentiation of adjacent soft tissues. A novel MRI technique called Sweep Imaging with Fourier Transformation (SWIFT) appears to be a suitable tool to overcome this challenge. The main advantage of SWIFT is to obtain signal from the cortical bone. We believe that the SWIFT technique will overcome the false positive results.

Patients enrolled in this study will be asked to come to the Center for Magnetic Resonance Research (CMRR) at the University of Minnesota, Minneapolis, Minnesota for a scheduled MRI. Brief scans will be obtained (less than 1 minute) to localize the area of interest. Longer MRI scans (around 5-15 minutes each) will then be obtained. The total time required for scanning will be about 1 hour.

To determine how well our MR images will predict the presence of mandibular invasion, we will compare our results with clinical, operative, radiological and pathological findings. Thus, patients will be asked to give permission to the investigators to access the relevant medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of oral cancer with clinical or imaging findings suggestive of maxillofacial or mandibular bone invasion.
* Patients who will be undergoing surgery as treatment for their oral cancer.

Exclusion Criteria:

* Pregnancy
* Ferromagnetic implant
* History of shotgun wounds and shrapnel
* Obesity (>250 pounds)
* Cardiac pacemaker
* MR incompatible medical device
* Severe claustrophobia
* Surgeries with potential ferromagnetic implants
* Metallic ink tattoo in close proximity to area of interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of oral cancer with clinical or imaging findings suggestive of maxillofacial or mandibular bone invation
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-04; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Ability of the newly created coil to detect mandibular bone invation in patients with squamous cell carcinoma adjacent to, or involving, the mandible. Comparison will be made to histopathological sections as the "gold standard". | Up to 15 months
  The goal of this outcome measure is to generate images, the quality of which are similar to histopathologic sections, with SWIFT MRI allowing determination of the presence or absence and degree of mandibular invasion of squamous cell carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Khariwala, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT01817140/Prot_SAP_000.pdf